CLINICAL TRIAL: NCT05406310
Title: Clinical Outcomes of Persistent Atrial Fibrillation Ablation Using Ablation Index-guided Radiofrequency Catheter Ablation in Patients With Continuous Monitoring
Acronym: AF-FAIR-MONTOR
Status: Withdrawn | Type: Observational
Why Stopped: Investigator left institution and did not transfer study to another institution or PI
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Other Study IDs: 32462
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Ablation; Ablation Index; Loop Recorder; Recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Ablation-Index guided ablation group: This is the prospective study group that will undergo persistent atrial fibrillation ablation guided by Ablation Index.
  Interventions: Device: Ablation Index-guided ablation
- High-power, short-duration ablation Group: This is another prospective group of patients who will undergo persistent atrial fibrillation ablation by high-power, short-duration using QDOT Micro catheter.
  Interventions: Device: High-power, short-duration ablation using QDOT Micro catheter

INTERVENTIONS:
Device: Ablation Index-guided ablation — Radiofrequency catheter ablation guided by Ablation Index software.
  Groups: Ablation-Index guided ablation group
Device: High-power, short-duration ablation using QDOT Micro catheter — Radiofrequency catheter ablation guided by high-power, short-duration ablation using QDOT Micro catheter
  Groups: High-power, short-duration ablation Group

SUMMARY:
Atrial fibrillation (AF) is the commonest condition affecting the rhythm of the heart. Tablets to try to normalize the heart rhythm rarely work well. As a result, doctors have devised a treatment called catheter ablation in which special wires are used to deliver heat energy (called ablation lesions) on the inside surface of the heart. Unfortunately, in many patients (almost 1 in 2), some of these ablation lesions recover, and that leads to the recurrence of AF. Many of these patients then need a second procedure to deliver further ablation at these recovered areas.

Because of that problem, a software called Ablation Index has been developed to optimize the delivery of ablation lesions. The study aims to find out the effectiveness of the use of that Ablation Index in improving the ablation outcomes in patients with persistent AF. Also, the study will test the effectiveness of a new ablation approach using a catheter which is capable of delivering high-power during ablation and therefore requires shorter time for ablation. This will be achieved by following up patients who received ablation for 12 months to monitor their response to treatment in terms of freedom from AF.

This study will include patients with persistent AF which means AF episode(s) that last for longer than seven days. Patients participating in the study will undergo their ablation treatment either guided by ablation Index or delivered using high-power, short-duration (HPSD) ablation.

All participants will undergo implantation of a cardiac monitor, also knowns as loop recorder, to monitor for recurrence of atrial tachyarrhythmia following ablation. The monitor stores these ECG recordings which will be downloaded during review appointments that will be arranged 6 weeks, 3 months, 6 months and 12 months after the ablation procedure.

All participants will undergo implantation of a cardiac monitor, also knowns as a loop recorder, to monitor for recurrence of atrial tachyarrhythmia following ablation. The monitor stores these ECG recordings which will be downloaded during review appointments that will be arranged 6 weeks, 3 months, 6 months, and 12 months after the ablation procedure.

DETAILED DESCRIPTION:
Single-center, prospective cohort study including patients with persistent AF (PeAF).

Primary Hypothesis:

Single AF ablation procedure that includes PVI achieved with point-by-point Wide Area Circumferential catheter ablation (WACA) either guided by Ablation Index (AI) targets or by HPSD ablation delivered using QDOT Micro catheter results in reduction in ATA as detected by insertable cardiac monitor (ICM).

Secondary hypotheses:

Single AF ablation procedure that includes PVI achieved with point-by-point WACA guided by Ablation Index targets has low incidence of adverse events and results in freedom from ATA, and improvement of AF symptoms and quality of life.

AF ablation procedures done by HPSD ablation delivered using QDOT Micro catheter will have shorter time and similar outcomes to procedures done using SmartTouch SF catheter guided by Ablation Index targets.

ELIGIBILITY:
Inclusion criteria:

* Aged over 18 years
* Persistent AF defined according to the 2017 HRS/EHRA/ECAS/APHRS/SOLAECE Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation, as AF episode that lasts longer than 7 days. (Calkins et al., 2017)
* Symptomatic despite drug treatment.
* Due to undergo AF ablation.

Exclusion criteria:

* Inability or unwillingness to receive oral anticoagulation with a Vitamin K antagonist (VKA) or non-VKA (NOAC) agent
* Previous catheter or surgical ablation procedure for AF
* Unwillingness or inability to complete the required follow-up arrangements
* Current pattern of paroxysmal AF
* Long standing persistent AF (continuous AF longer than 12 months before ablation)
* Prior prosthetic mitral valve replacement or severe structural cardiac abnormality
* Known infiltrative cardiomyopathy
* Known severe left ventricular systolic function (ejection fraction <35%)
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persistent atrial fibrillation patients who are 18 years or older and are indicated for atrial fibrillation ablation and have no exclusion criteria as listed above.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
ICM-detected ATA burden | 12 months
  ICM-detected ATA burden measured as percentage of time spent in ATA (i.e., hours of ATA/hours of monitoring X 100)

SECONDARY OUTCOMES:
The occurrence of ATA recurrence of 2 minutes or more | 12 month
QOL | 6 and 12 months after initial ablation
  QOL 6 and 12 months after initial ablation, as quantified by the validated AFEQT questionnaire.
Major complication rates | Within 60 days after a PVI procedure
  Major complications include cardiac tamponade, stroke/TIA, myocardial infarction, phrenic nerve paralysis, oesophageal perforation/atrio-oesophageal fistula, major vascular complications, and death.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hussein A, Das M, Riva S, Morgan M, Ronayne C, Sahni A, Shaw M, Todd D, Hall M, Modi S, Natale A, Dello Russo A, Snowdon R, Gupta D. Use of Ablation Index-Guided Ablation Results in High Rates of Durable Pulmonary Vein Isolation and Freedom From Arrhythmia in Persistent Atrial Fibrillation Patients: The PRAISE Study Results. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006576. doi: 10.1161/CIRCEP.118.006576. PMID 30354288
- [Background] Hussein A, Das M, Chaturvedi V, Asfour IK, Daryanani N, Morgan M, Ronayne C, Shaw M, Snowdon R, Gupta D. Prospective use of Ablation Index targets improves clinical outcomes following ablation for atrial fibrillation. J Cardiovasc Electrophysiol. 2017 Sep;28(9):1037-1047. doi: 10.1111/jce.13281. Epub 2017 Jul 26. PMID 28639728